CLINICAL TRIAL: NCT05036330
Title: ProvoxLife® Adoption Trends for Heat-Moisture Exchanger (HME): The PATH Registry
Brief Title: ProvoxLife Adoption Trends for Heat-Moisture Exchanger
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2020-1114; NCI-2021-08784 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1114 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-08-25; First posted 2021-09-05 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Malignant Head and Neck Neoplasm
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (evaluation, examination, questionnaire): Patients undergo speech and swallow evaluation by speech pathologist or study staff member and examination of TEP and laryngectomy stoma. Patients also complete questionnaires over 30 minutes about use the ProvoxLife HME system, symptoms, ability to communicate, exercise and physical activity levels, and quality of life at baseline and 3 months post-ProvoxLife.
  Interventions: Other: Clinical Evaluation; Procedure: Physical Examination; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Clinical Evaluation — Undergo speech and swallow evaluation
  Other Names: Clinical Assessment
Procedure: Physical Examination — Undergo examination of TEP and laryngectomy stoma
  Other Names: Assessment; General Examination
Other: Quality-of-Life Assessment — Complete questionnaires
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study examines factors that affect how often patients who have a total laryngectomy use a ProvoxLife heat-moisture exchanger (HME) system to help improve their lung function. ProvoxLife HMEs are single use heat- and moisture exchangers for patients breathing through a tracheostoma. Information from this study may help doctors learn more about factors associated with patterns of use and how often patients use the ProvoxLife HME system.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine clinical and patient factors associated with patterns of use of the ProvoxLife HME system for pulmonary rehabilitation after total laryngectomy.

SECONDARY OBJECTIVES:

I. To explore outcomes associated with patterns of ProvoxLife HME system. II. To explore factors associated with post-laryngectomy outcomes.

OUTLINE:

Patients undergo speech and swallow evaluation by speech pathologist or study staff member and examination of tracheoesophageal puncture (TEP) and laryngectomy stoma. Patients also complete questionnaires over 30 minutes about use the ProvoxLife HME system, symptoms, ability to communicate, exercise and physical activity levels, and quality of life at baseline and 3 months post-ProvoxLife.

ELIGIBILITY:
Inclusion Criteria:

* Adults >= 18 years of age planned for or status post total laryngectomy
* Using or ready for fit of HME system

Exclusion Criteria:

* Active malignancy if post-total laryngectomy (TL) at the time of enrollment
* Unable to complete questionnaires in English language

  * The primary endpoint derives from a study specific questionnaire, due to limited resources, is only available in English language
* Cognitive or other limitations that preclude independent self-care or completion of questionnaires

  * Cognitive or other limitations that preclude independent self-care or completion of questionnaires will be assessed in the screening interview by the clinical or research team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients using or planning to use HME as part of standard care
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
To determine clinical and patient factors associated with patterns of use of the ProvoxLife HME system for pulmonary rehabilitation after total laryngectomy. | Up to 3 months post-ProvoxLife HME

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A Hutcheson, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org